CLINICAL TRIAL: NCT01672541
Title: Randomized Controlled Trial of the "Dating Matters: Strategies to Promote Healthy Teen Relationships" Comprehensive Approach
Brief Title: Dating Matters: Strategies to Promote Healthy Teen Relationships
Acronym: DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: NORC at the University of Chicago (Other); Ogilvy Public Relations (Unknown); Alameda County Public Health Department (Unknown); Baltimore City Health Department (Other); Broward County Health Department (Unknown); Chicago Department of Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCIPC-6161
Record Dates: First submitted 2012-08-20; First posted 2012-08-27 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2018-01

CONDITIONS: Teen Dating Violence; Healthy Dating Relationship Behaviors
Keywords: dating violence; healthy relationship behaviors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dating Matters Comprehensive Approach (Experimental): Schools randomly assigned to the comprehensive approach will: implement 6th, 7th, and 8th grade student curricula in English to all the students in these grades; offer parent programs for parents of 6th, 7th, and 8th graders;implement a communications campaign involving brand ambassadors, a text message campaign, and social media campaign;encourage all educators to take an online training about teen dating violence for educators;be supported in assessing and informing local school or community policies relevant to teen dating violence.
  Interventions: Behavioral: Dating Matters Comprehensive Approach
- Standard of Care Safe Dates Approach (Active Comparator): Schools randomly assigned to the standard of care approach will implement Safe Dates as it is published in their schools 8th grade classes.
  Interventions: Behavioral: Standard of Care Safe Dates Approach

INTERVENTIONS:
Behavioral: Dating Matters Comprehensive Approach — The Dating Matters Comprehensive Approach includes:
  6th, 7th, and 8th grade Student Curricula; Parent Programs for parents of 6th, 7th, and 8th graders; A communications campaign involving brand ambassadors, a text message campaign, and social media campaign; An online training about teen dating violence for educators; Developmental component: A guidance document for sites on assessing and informing local policies relevant to teen dating violence for comprehensive schools (likely to be substantial cross and within site variation on this component)
  Arms: Dating Matters Comprehensive Approach
Behavioral: Standard of Care Safe Dates Approach — Safe Dates curriculum for 8th grade students
  Arms: Standard of Care Safe Dates Approach

SUMMARY:
The Dating Matters: Strategies to Promote Healthy Teen Relationships Initiative intends to promote respectful, nonviolent dating relationships among adolescents living in high-risk, urban communities. CDC has developed a comprehensive approach to promoting respectful, non-violent relationships based on current evidence based and evidence informed strategies. This comprehensive approach includes: school-based curricula for 6th, 7th, and 8th grade students; separate parent programs for parents of 6th, 7th, and 8th grade students; a communications campaign involving social media and near-peer brand ambassadors; an online training about dating violence for educators; policy assessment at the school or community level; and development and validation of school and community level indicators of teen dating violence. Additionally, schools assigned to the comprehensive condition will also receive intensive training and technical assistance to support implementation of these components. Among 4 U.S. sites, 44 schools will be randomly assigned to implement either the Dating Matters comprehensive approach or the "standard of care" approach, which we are operationalizing as Safe Dates, a an evidence based student curriculum for 8th graders. We hypothesize that the comprehensive approach will be more effective than the standard approach at preventing the perpetration and victimization of teen dating violence over time and at promoting positive relationship behaviors over time.

DETAILED DESCRIPTION:
Dating Matters: Strategies to Promote Healthy Teen Relationships Initiative is intended to promote respectful, nonviolent dating relationships among adolescents living in high-risk, urban communities. The objective of this project is to develop, implement, and evaluate a comprehensive approach to promoting respectful, nonviolent teen dating relationships by utilizing current evidence-based practice and experience. The focus on high-risk, urban communities is predicated on data that suggest that the prevalence of dating violence among middle school students is higher in urban communities (O'Leary & Slep, in press). Moreover, this project aims to fill a gap in our understanding of teen dating violence (TDV) prevention because existing effective TDV prevention programs have not been identified for these high-risk settings.

CDC's comprehensive approach, the Dating Matters: Strategies to Promote Healthy Teen Relationships Initiative, includes components at multiple ecological domains, individual level, family-level and broader school/community level. Specifically, the initiative includes: (1) school-based implementation of a CDC-developed healthy relationship curriculum in the 6th and 7th grade and an adaptation of an evidence based TDV curriculum (Safe Dates) in the 8th grade; (2) implementation of a 6th (Parents Matter with added TDV content), 7th (CDC developed), and 8th (Families for Safe Dates) grade parent-curriculum; (3) an on-going communications campaign implemented throughout the initiative, which includes a Brand Ambassador adolescent program; (4) educator completion of an online training on the risk factors and warning signs of TDV; (5) policy assessment and information at a school or community level; and, (6) development and validation of school and community-level indicators of TDV. In addition to these components, the schools implementing Dating Matters will also receive additional training and technical assistance in adapting these programs with surface level adaptations to make them more culturally relevant to their specific populations.

CDC is funding the local, city, or county public health departments in Chicago, Illinois, Alameda County (Oakland), California, Broward County (Ft. Lauderdale), Florida, and Baltimore, Maryland to implement the two models of TDV prevention that will be evaluated in the outcome and implementation evaluation: the comprehensive Dating Matters initiative and the standard of care model, which is Safe Dates implemented in 8th grade. These health departments collectively have identified 44 schools in high-risk urban communities; we have randomly assigned half the schools to implement the comprehensive model with intensive technical assistance and half to implement the standard of care model with basic technical assistance. These sites were awarded September 13, 2011.

The purpose of the trial is to determine the effectiveness of the comprehensive approach (Dating Matters) compared with standard practice in TDV prevention (Safe Dates only implemented in 8th grade). Outcome measures for determining effectiveness will be derived primarily from surveys with students, parents, and school educators. However, in addition to surveys, we will also be conducting focus groups with students, curriculum implementers, and brand ambassasors, as well as surveys with brand ambassadors, as sources of process, rather than outcome, measures. These process measures may be used to improve program fidelity, improve program components, or as factors in outcome analyses.

ELIGIBILITY:
Inclusion Criteria:

* Students, parents, and educators at the schools identified for participation in the study

Exclusion Criteria:

* Students and educators must be able to participate in interventions and complete surveys in English: Parents must be able to participate in interventions and complete surveys in English or Spanish. Those not able to do this due to languages spoken will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10000 (Actual)
Dates: Start 2012-08; Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Perpetration of dating violence | 2 times per year for up to 6 years
  Student self-report of perpetration of physical, sexual, and psychological violence and/or stalking against a dating partner
Victimization of dating violence | 2 times per year for up to 6 years
  Student self- report of victimization of physical, sexual, and psychological violence and/or stalking from a dating partner
Engagement in healthy relationship behaviors | 2 times per year for up to 6 years
  Student self-report of engagement in healthy relationship behaviors (i.e., good communication, conflict management, etc) with a dating partner

SECONDARY OUTCOMES:
Attitudes toward the acceptability of dating violence | 2 times per year for up to 6 years
  Student self report of attitudes toward TDV; Parent self report of attitudes toward TDV; Educator report of students's attitudes toward TDV (2x/year the first year, 1x/year after that)
Knowledge about teen dating violence | 2 times per year for up to 6 years
  Student self report of knowledge of facts about TDV; Parent self report of knowledge of facts about TDV
Attitudes toward gender roles | 2 times per year for up to 6 years
  Student self-report of attitudes toward male and female gender roles (2x/year through 12th grade, so up to 6 years for those who start the study in 6th grade) Parent self-report of attitudes toward male and female gender roles (2x/year for up to 3 years)
Knowledge Regarding Available Resources | 2 times per year for up to 6 years
  Student self-report of awareness of community and national resources for helping teenagers in abusive and violent relationships
Positive parenting behaviors | 2 times per year, for up to 6 years
  Student report of of parent's engagement in positive parenting behaviors, such as praise; of parental monitoring of dating (e.g., parent knows the people the student dates); of general parental monitoring behaviors (e.g., parent knows where student goes out at night) (up to 6 years); Parent report of: of general monitoring behaviors; of monitoring of child's dating; of engagement in positive parenting behaviors toward child; of involvement in child's life and activities, of use of positive discipline techniques toward the child, of use of corporal punishment of the child, and of consistency of discipline toward the child (up to 3 years)
Perpetration of sexual harassment | 2 times per year for up to 6 years
  Student self report of engagement in sexual harassment behaviors toward others, in person and online
Victimization of sexual harassment | 2 times per year for up to 6 years
  Student self report of victimization of sexual harrasment by others, in person and online
School climate | 2 times per year for up to 6 years
  Student report of school climate and safety (2x/ year up to 6 years); Educator report of school climate and safety (2x/year first year, 1x per year after); Student self-report of social support from a teacher or other adult in school
Engagement in risky behaviors | 2 times per year for up to 6 years
  Student self report of engagement in risky behaviors such as risky sex, substance use, aggression, and delinquency
Student mental health | 2 times per year for up to 6 years
  Student self-report of depressive and anxious symptomology.
Student prosocial behaivor | 2 times per year for up to 6 years
  Student self report of engagment in prosocial behavior such as helping others, sharing.
Parental attitudes toward and rules about dating | 2 times per year for up to 3 years
  Parent report about their attitudes toward their child dating, any rules they have for their child about dating, and their communication with their child about those rules
Parent-child communication about risk behaviors | 2 times per year for up to 3 years
  Parent report about the extent to which parent and child communicate about topics such as dating, drugs, sex and sexually transmitted infections
Parent relationship quality | 2 times per year for up to 3 years
  Parent report on communication and satisfaction with communication between him or her and his or her partner Parent self-report of satisfaction with relationship with partner
Parent engagement in Intimate Partner Violence (IPV) | 2 times per year for up to 3 years
  Parent report of perpetration or victimization of IPV
Dating Violence and sexual harassment visibility in school | 2 times per year first year, 1 time per year for 3 more years
  Educator self-report of witnessing dating violence and seuxal harassment in thie school.
Educator ability to address teen dating violence | 2 times per year first year, 1 time per year for 3 more years
  Educator report of views toward teen dating violence prevention and confidence in discussing the issue with students Educator report of knowledge of and responsibility to intervene when witnessing teen dating violence and harassment
Issues faced by youth | 2 times per year first year, 1 time per year for 3 more years
  Educator report of the most common issues (e.g., drugs) faced by students in the school
Parent ability to detect TDV | 2 times per year for up to 3 years
  Parent self-report in confidence in ability to detect teen dating violence perpetration and victimization in child
Exposure to the communications campaign | 2 times per year for up to 6 years
  Student self-report of awareness of the communication campaign, including whether the student has heard of and participated in the i2i campaign activities.

OTHER OUTCOMES:
Demographic variables | 2 times per year for up to 6 years
  * Student self-report of demographic factors, such as age, gender, race/ethnicity, household composition, and relationship history;
  * Parent self-report of demographic factors, such as age, gender, race/ethnicity, household composition, total family income, educational attainment, and relationship history;
  * Educator self-report of demographic factors, such as race/ethnicity and gender
Experience delivering prevention programs | 2 times per year first year, 1 time per year for 3 more years
  Educator self-report of experience delivering prevention programs, such as teen dating violence and harassment prevention programs
Religiosity | 2 times per year for up to 3 years
  Parent self-report of attendance at religious services and importance of religious beliefs
Student extra curricular activities | 2 times per year for up to 3 years
  Parent report of student engagement in extra-curricular activities
Housing stability | 2 times per year for up to 3 years
  Parent report of stability of housing for both parent and student (e.g., how long lived in the same neighborhood)
Neighborhood cohesion | 2 times per year for up to 3 years
  Parent report of characteristics of the neighborhood, such as the extent to which individuals in the neighborhood would intervene if a youth needed help and/or was engaging in delinquent behavior
Gang involvement | 2 times per year for up to 6 years
  Student self report of having been initiated into a gang
Exposure to intimate partner violence | 2 times per year for up to 6 years
  Student self-report of witnessed (by seeing or hearing) intimate partner violence between a parent/guardian and his/her partner
Exposure to community violence | 2 times per year for up to 6 years
  Student self-report of witnessed (by seeing or hearing) community violence, such as hearing or seeing gun shots or others being physically attacked
Views toward Dating Matters sustainability | 2 times per year first year, 1 time per year for 3 more years
  Educator report of views regarding Dating Matters sustainability, including level of commitment to sustainability

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis H Niolon, Ph.D., Principal Investigator — Centers for Disease Control and Prevention
Locations (4):
- United States (4):
  - Alameda County Public Health Department, Oakland, California
  - Broward County Health Department, Fort Lauderdale, Florida
  - Chicago Department of Public Health, Chicago, Illinois
  - Baltimore City Health Department, Baltimore, Maryland

REFERENCES:
- [Derived] Niolon PH, Estefan LF, DeGue S, Le VD, Tracy AJ, Ray C, Bontempo D, Little TD, Vivolo-Kantor AM, Latzman N, Taylor B, Tharp A. High School Follow-Up of the Dating Matters(R) RCT: Effects on Teen Dating Violence and Relationship Behaviors. Prev Sci. 2024 May;25(4):603-615. doi: 10.1007/s11121-024-01648-z. Epub 2024 Mar 8. PMID 38459353
- [Derived] Espelage DL, Rulison KL, Ingram KM, Valido A, Schmeelk-Cone K, Wyman PA. Social Networks of Adolescent Sexual Violence Perpetrators: Peer Friendship and Trusted Adult Characteristics. Prev Sci. 2022 Jan;23(1):154-166. doi: 10.1007/s11121-021-01296-7. Epub 2021 Sep 3. PMID 34480329
- [Derived] DeGue S, Niolon PH, Estefan LF, Tracy AJ, Le VD, Vivolo-Kantor AM, Little TD, Latzman NE, Tharp A, Lang KM, Taylor B. Effects of Dating Matters(R) on Sexual Violence and Sexual Harassment Outcomes among Middle School Youth: a Cluster-Randomized Controlled Trial. Prev Sci. 2021 Feb;22(2):175-185. doi: 10.1007/s11121-020-01152-0. PMID 32844328
- [Derived] Estefan LF, Vivolo-Kantor AM, Niolon PH, Le VD, Tracy AJ, Little TD, DeGue S, Latzman NE, Tharp A, Lang KM, McIntosh WL. Effects of the Dating Matters(R) Comprehensive Prevention Model on Health- and Delinquency-Related Risk Behaviors in Middle School Youth: a Cluster-Randomized Controlled Trial. Prev Sci. 2021 Feb;22(2):163-174. doi: 10.1007/s11121-020-01114-6. PMID 32242288
- [Derived] Vivolo-Kantor AM, Niolon PH, Estefan LF, Le VD, Tracy AJ, Latzman NE, Little TD, Lang KM, DeGue S, Tharp AT. Middle School Effects of the Dating Matters(R) Comprehensive Teen Dating Violence Prevention Model on Physical Violence, Bullying, and Cyberbullying: a Cluster-Randomized Controlled Trial. Prev Sci. 2021 Feb;22(2):151-161. doi: 10.1007/s11121-019-01071-9. PMID 31833020
- [Derived] Niolon PH, Vivolo-Kantor AM, Tracy AJ, Latzman NE, Little TD, DeGue S, Lang KM, Estefan LF, Ghazarian SR, McIntosh WLK, Taylor B, Johnson LL, Kuoh H, Burton T, Fortson B, Mumford EA, Nelson SC, Joseph H, Valle LA, Tharp AT. An RCT of Dating Matters: Effects on Teen Dating Violence and Relationship Behaviors. Am J Prev Med. 2019 Jul;57(1):13-23. doi: 10.1016/j.amepre.2019.02.022. Epub 2019 May 22. PMID 31128957